CLINICAL TRIAL: NCT01488331
Title: A Patient Cohort With Locally Advanced or Metastatic Non-small Cell Lung Cancer Treated With Tarceva (Erlotinib) Monotherapy and Not Progressing After at Least 9 Months
Brief Title: An Observational Study of Tarceva (Erlotinib) in Patients With Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22973
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multi-center, observational study will assess the progression-free survival and safety of patients with locally advanced or metastatic non-small cell lung cancer treated with Tarceva (erlotinib) and not disease progressing after at least 9 months. Data will be collected for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of locally advanced or metastatic non-small cell lung cancer (NSCLC, stage III/IV)
* Treatment with Tarceva monotherapy and not progressing after at least 9 months at the date of study start

Exclusion Criteria:

* Not agreeing to be followed-up (for a maximum of 24 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 24 months

SECONDARY OUTCOMES:
Best treatment response | 24 months
Overall survival | 24 months
Safety (incidence of adverse events) | 24 months
Type of treatment response | 24 months
Treatment compliance of patient | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (81):
- France (81):
  - Abbeville
  - Agen
  - Aix-en-Provence
  - Ajaccio
  - Amiens
  - Angers
  - Annecy
  - Aubagne
  - Auxerre
  - Bastia
  - Bordeaux
  - Bourg-en-Bresse
  - Brest
  - Bron
  - Bry-sur-Marne
  - Caen
  - Cagnes-sur-Mer
  - Chalon-sur-Saône
  - Chambray-lès-Tours
  - Chaumont
  - Chauny
  - Cholet
  - Clamart
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Coquelles
  - Cornebarrieu
  - Creil
  - Créteil
  - Dax
  - Dijon
  - Draguignan
  - Eaubonne
  - Fréjus
  - Gap
  - Gleizé
  - Helfaut
  - Hyères
  - La Chaussée-Saint-Victor
  - La Roche-sur-Yon
  - La Rochelle
  - La Source
  - La Tronche
  - Le Plessis-Robinson
  - Libourne
  - Limoges
  - Longjumeau
  - Lyon
  - Meaux
  - Metz
  - Meudon
  - Montauban
  - Montpellier
  - Mulhouse
  - Nancy
  - Nantes
  - Nevers
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Pontoise
  - Reims
  - Rennes
  - Rouen
  - Saint-Aubin-lès-Elbeuf
  - Saint-Avold
  - Saint-Brieuc
  - Saint-Jean
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Salon-de-Provence
  - Senlis
  - Strasbourg
  - Tarbes
  - Thionville
  - Toulon
  - Toulouse
  - Tours
  - Vénissieux
  - Vichy